CLINICAL TRIAL: NCT02237261
Title: Bendamustine, Prednisone and Velcade® for First-line Treatment of Patients With Symptomatic Multiple Myeloma Not Eligible for High-dose Chemotherapy Followed by Autologous Stem Cell Transplantation (BPV).
Brief Title: Bendamustine, Prednisone and Velcade® for First-line Treatment of Patients With Symptomatic Multiple Myeloma
Acronym: BPV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: German Cancer Research Center (Other); Janssen-Cilag International NV (Industry); Mundipharma Research GmbH & Co KG (Industry); inVentiv Health Clinical (Other)
Responsible Party: Principal Investigator, Dr. Marc Raab, Marc S. Raab MD, Medical Hospital V (Hematology, Oncology, Rheumatology), Section multiple myeloma, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV; 2013-005485-19 (EudraCT Number)
Record Dates: First submitted 2014-06-09; First posted 2014-09-11 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Multiple Myeloma
Keywords: Newly diagnosed symptomatic multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; Bortezomib; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine, Bortezomib, Prednisone (Experimental): Induction: Bortezomib: 1.3 mg/m2 subcutaneous for 7 days and Bendamustine: 90 mg/m2 intravenous for 2 days and in addition Prednison: : 60 mg/m2 per os for 4 days Consolidation: Bortezomib: 1.3 mg/m2 subcutaneous for 4 days and Bendamustine: 90 mg/m2 intravenous for 2 days and in addition Prednison 60 mg/m2 per os for 4 days
  Interventions: Drug: Bendamustine, Bortezomib, Prednisone

INTERVENTIONS:
Drug: Bendamustine, Bortezomib, Prednisone — Cycle 1 (d1-42) - Induction:
  Bortezomib: 1.3 mg/m2 s.c.: d1, 4, 8, 11, 22, 25, 29, 32 Bendamustine: 90 mg/m2 iv, d1, 2 Prednison: : 60 mg/m2 po,, d1-4
  Cycle 2-9 (d1-28) - Consolidation:
  Bortezomib: 1.3 mg/m2 s.c.: d1, 8, 15, 22 Bendamustine: 90 mg/m2 iv: d1, 2 Prednison: 60 mg/m2 po: d1-4
  Other Names: Velcade (Bortezomib); Levact (Bendamustine)

SUMMARY:
The purpose of this study is to improve efficacy of treatment for patients with newly diagnosed multiple myeloma who are not eligible for high-dose chemotherapy followed by autologous stem cell transplantation by Bendamustin, Bortezomib (Velcade), and Prednisone.

DETAILED DESCRIPTION:
1. Objectives Primary

   -Therapeutic efficacy of BPV regimen for multiple myeloma as evidenced by the overall response defined as partial response (PR) or better

   Secondary
   * to assess overall survival (OS) and progression-free survival (PFS)
   * to determine response duration
   * to investigate improvements of renal function
   * to evaluate safety and toxicity (with respect to adverse events of CTCAE grade ≧3 and SAEs)
   * to analyze the efficacy for genetically defined subgroups of myeloma patients based on iFISH and gene-expression profiling
2. Investigational Medicinal Products Bortezomib Bendamustine both in combination with Prednisone

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed multiple myeloma requiring systemic treatment (according to CRAB criteria as specified in the appendix I) with following characteristics: Subject is not a candidate for high-dose chemotherapy and stem cell transplantation due to age, presence of comorbidities likely to have a negative impact on tolerability of HDT-SCT, or subject preference
2. Measurable disease, defined as any quantifiable monoclonal protein value, defined by at least one of the following three measurements (Durie et al., 2006):

   * Serum M-protein ≥ 10g/l
   * Urine light-chain (M-protein) of ≥ 200 mg/24 hours
   * Serum FLC assay: involved FLC level ≥ 10 mg/dl provided sFLC ratio is abnormal
3. Age>18 years
4. WHO performance status 0-3 (WHO=3 is allowed only when related to MM and not to co-morbid conditions) (see appendix III)
5. For women of childbearing potential: negative pregnancy test at inclusion
6. All patients must be willing and capable to use adequate contraception during the complete therapy.
7. All patients must agree to abstain from donating blood while on study
8. Ability to understand character and individual consequences of the clinical trial
9. Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* Subjects presenting any of the following criteria will not be included in the trial

  1. Patient has known hypersensitivity to bortezomib, bendamustine and prednisone or to any of the constituent compounds (incl. boron and mannitol).
  2. Systemic AL amyloidosis (except for patients with AL amyloidosis of the skin or the bone marrow)
  3. Chemotherapy or radiotherapy during the past 5 years except patients with local radiotherapy in case of local myeloma progression. (Note: patients may have received a cumulative dose of up to 160 mg of dexamethasone or equivalent as emergency therapy within 3 weeks prior to study entry.)
  4. Plasma cell leukemia which requires the presence of 20% of plasma cell in peripheral blood leukocytes and at least 2 plasma cells/nl.
  5. Severe cardiac dysfunction (NYHA classification III-IV, see appendix III)
  6. Significant hepatic dysfunction (serum bilirubin ≥ 2 mg/dl or ASAT and/or ALAT ≥ 2.5 times normal level), unless related to myeloma
  7. Patients known to be HIV-positive
  8. Patients with active, uncontrolled infections
  9. Patients with peripheral neuropathy or neuropathic pain of CTC grade 2 or higher (as defined by the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0, see appendix V)
  10. Second malignancy during the past 5 years except:
* Adequately treated basal cell or squamous cell skin cancer, or
* Carcinoma in situ of the cervix, or
* Prostate cancer < Gleason score 6 with undetectable prostate-specific antigen (PSA) over 12 months, or
* Ductal breast carcinoma in situ with full surgical resection (i.e., negative margins), or
* Similar malignant condition as a.- d. with an expected5-year disease free survival larger than 95% 11. Patients with acute diffuse infiltrative pulmonary and pericardial disease 12. Autoimmune hemolytic anemia with positive Coombs test or immune thrombocytopenia 13. Platelet count < 50 x 109/l (transfusion support within 14 days before the test is not allowed), unless related to myeloma 14. Hemoglobin < 7.5g/dl, unless related to myeloma 15. Absolute neutrophil count (ANC) < 0.75 x 109/l (the use of colony stimulating factors within 14 days before the test is not allowed), unless related to myeloma 16. Pregnancy and lactation 17. Participation in other clinical trials within one month prior to enrolment except for supportive care studies and vaccination studies. (Note: this does not include long-term follow-up periods without active drug treatment of previous studies during the last 6 months).

No subject will be allowed to enrol in this trial more than once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) of BPV | 2 years
  ORR is defined as PR or better

SECONDARY OUTCOMES:
Number and percentage of patients achieving a complete response | 2 years
  Number and percentage of patients achieving a complete response
Progression-free survival (PFS) | 2 years
  PFS defined as time from registration to progression or death whatever comes first
Overall survival (OS) | 2 years
  OS defined as time from registration to time of death from any cause.
Time-to-progression (TTP) | 2 years
  TTP defined as time from registration to disease progression. TTP is censored at time of deaths which are not caused by progression.
Disease-free survival (DFS) | 2 years
  DFS defined as time from start of CR to relapse or death from any cause whichever comes first. Patients evaluable for DFS are patients in complete Response.
Duration of response (DOR) | 2 years
  DOR defined as time from first observation of PR to the time of disease progression.
Renal response according to IMWG (CRrenal, PRrenal, MRrenal) | 2 years
  percent of patients with recovery/improvement of renal function (for patients with impared renal finction at baseline)
Toxicity (with respect to adverse events of CTCAE grade ≧3 and SAEs) | 2 years
  toxicity during study therapy with AE of CTC grade ≧ 3, as well as neuropathy of CTC grade 2, measured by CTC-AE (v4.0).
Time to objective Response (TOR) | 2 years
  TOR defined as time from registration to achieving an objective response for patients achieving an objective Response.
Time to treatment failure (TTF) | 2 years
  TTF is defined as time from registration to treatment discontinuation for any reason, including disease progression, Treatment toxicity, patient preference or death.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Knauf, MD, Study Chair — Hematology/Oncology,Bethanien hospital, Im Pruefling 17-19, 60389 Frankfurt/M., Germany
Locations (15):
- Germany (15):
  - Mannheimer Onkologie Praxis, Mannheim, Ba-Wü
  - Onkologische Schwerpunktpraxis, Heidelberg, Baden-Wurttemberg
  - Medizinische Klinik V, Universitätsklinikum Heidelberg, Sektion Multiples Myelom, Heidelberg, Baden-Wurttemberg
  - Hämatologisch-Onkologische gemeinschaftspraxis, Augsburg, Bavaria
  - Gemeinschaftspraxis Dr. R. Schlag/Dr. B. Schöttker, Würzburg, Bavaria
  - Onkologische Schwerpunktpraxis Dr. G. Kojouharoff, Darmstadt, Hesse
  - Hämatologisch-Onkologische Gemeinschaftspraxis am Bethanienkrankenhaus, Frankfurt am Main, Hesse
  - Agaplesion Markus Krankenhaus gGmbH, Medizinisches Versorgungszentrum, Frankfurt am Main, Hesse
  - Onkologische Gemeinschaftspraxis, Cologne, North Rhine-Westphalia
  - Onkologisches Ambulanzzentrum Hannover am Diakoniekrankenhaus Henriettenstift gGmbH, Hannover, North Rhine-Westphalia
  - Klinikum Idar-Oberstein GmbH, Innere Medizin I, Idar-Oberstein, Rh-Pfalz
  - Onkologische Schwerpunktpraxis Speyer, Speyer, Rhineland-Palatinate
  - Städtische Klinikum Dessau, Dessau, Saxony-Anhalt
  - Klinikum Aschaffenburg, Med. Klinik II, Aschaffenburg
  - Onkologische Praxis Oldenburg/Delmenhorst, Oldenburg

REFERENCES:
- [Result] Knauf W, Dingeldein G, Schlag R, Welslau M, Moehler T, Terzer T, Walter S, Habermehl C, Kunz C, Goldschmidt H, Raab MS; BPV trial group. First-line therapy with bendamustine/prednisone/bortezomib-A GMMG trial for non-transplant eligible symptomatic multiple myeloma patients. Eur J Haematol. 2020 Aug;105(2):116-125. doi: 10.1111/ejh.13409. Epub 2020 May 26. PMID 32155662